CLINICAL TRIAL: NCT02069873
Title: Phase II Efficacy Study on Group Delivery of Effective Treatments for PTSD
Brief Title: Effectiveness of Cognitive, Exposure, and Skills Group Manualized Treatments in Operations Iraqi (OIF)/Operation Enduring Freedom (OEF) Female Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Diane T. Castillo, Ph.D., Supervisory Psychologist, New Mexico VA Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-08-2-0022; PT074309 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-02-14; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; Group; Treatment; Cognitive, Exposure, Skills; Women; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 16-Week Group Treatment (Experimental): The 16-week treatment group will contain 3 blocks of treatment (exposure, cognitive, skills) with order randomized within the treatment. The first and last group session are considered inactive treatment sessions. The group treatment will be provided weekly.
  Interventions: Behavioral: 16-Week Group Treatment
- Wait List Control (No Intervention): The Wait List Control group will receive minimal attention, as they will meet bi-monthly for supportive sessions with the study psychologist. The study psychologist will not introduce any active treatment in the individual sessions.

INTERVENTIONS:
Behavioral: 16-Week Group Treatment — Within the 16-week group treatment, the cognitive block will contain 5 sessions, the exposure block will contain 5 sessions, and the skills block will contain 4 sessions.
  Other Names: Cognitive treatment; Exposure treatment; Skills treatment; Group treatment
  Arms: 16-Week Group Treatment

SUMMARY:
The purpose of the study is to evaluate the efficacy of a group protocol for the delivery of evidence-based therapies in comparison to a wait-list control and evaluate the relative contribution of exposure, cognitive, and skills blocks of treatment in a 16-session manualized group treatment protocol in a sample of OIF/OEF female PTSD veterans. Hyp1: Overall improvement is expected in PTSD symptoms compared to a wait-list control group; and Hyp2: the exposure and cognitive components are expected to show greater improvement in PTSD symptoms than the skills component. Significant results will establish the efficacy of a group format for evidence-based treatments for all veterans with a PTSD diagnosis. An ancillary part of the study is to examine initial neuropsychological presentation in this population and possible changes that may occur as the result of treatment.

DETAILED DESCRIPTION:
OBJECTIVES: The objectives are to 1) evaluate the effectiveness of exposure, cognitive, and skills (assertiveness/relaxation) therapies within a 16-session group; and 2) evaluate the relative contribution of each of three treatment components in a manualized treatment group in a sample of OIF/OEF female PTSD veterans. HYPOTHESES: Hypothesis 1. Female OIF/OEF PTSD veterans will show reductions in PTSD symptoms and improvement in general functioning after participation in a structured group treatment compared to a wait-list control group. Hypothesis 2. Exposure and cognitive components will show greater improvement in PTSD symptoms than the skills component. RESEARCH DESIGN/BACKGROUND: Based on studies with male combat veterans, female civilian rape victims, and female veterans, therapies most effective for Posttraumatic Stress Disorder (PTSD) are exposure therapy (1,2,3) and cognitive restructuring (4), with less improvement found in other treatments, such as relaxation and assertiveness training (5). Most examinations of PTSD treatments have been conducted in an individual format, but most PTSD treatments offered in Veterans Administration (VA) hospital PTSD programs are conducted in a group format (6). It is critical to determine if these therapies work in a group setting, as only one study (7) found no differences in exposure therapy compared to a support group. In a comprehensive manualized group treatment protocol (8) exposure therapy provided in a group was found effective (9). The aim of the present study is to establish the effectiveness of exposure therapy, among other evidence-based therapies, in a well designed randomized study. METHODOLOGY: Castillo's (8) manualized group treatment protocol for female veterans with PTSD will be modified into a 16-week treatment group with a five-week exposure, five-week cognitive, and four-week skills treatment blocks. Seventy-two subjects will be assessed with structured interviews (SCID and CAPS) and questionnaires (Traumatic Life Events and Quality of Life Inventory) and randomized into one of two arms: 16-week immediate treatment, or a 16-week wait-list control, the latter of which will be reassessed and offered the study treatment. Oversampling will result in 72 subjects in the active treatment arm. Subjects will be reassessed upon completion of treatment or wait-list, at 3, and 6 months following treatment. All treatment groups will include three female OIF/OEF veterans positive for PTSD. The treatment blocks will be varied into six possible orders to control for order effects and the PTSD Symptom Checklist will be administered after each treatment block. Data will be collected for three years. CLINICAL RELATIONSHIPS: Significant results will contribute to the establishment of evidence-based treatments in a manualized treatment group for all veterans with a PTSD diagnosis. FINDINGS: Present findings from Dr. Castillo's lab suggest the effectiveness of exposure therapy in a group setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD
* Iraq or Afghanistan female Veteran
* Psychiatry stability (no suicide, homicide)
* One clear memory of a trauma
* Stability on psychiatric medications for 1 month

Exclusion Criteria:

* Active substance use/abuse (or in remission less than 3 mo)
* Psychotic symptoms or diagnosis
* Bipolar disorder diagnosis
* Cognitive impairment
* Involvement in a violent relationship
* Self mutilation within past 6 months

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in PTSD from baseline on the Clinician Administered PTSD Scale (CAPS) to post-treatment, 3 months, and 6 months later. | Baseline, post-treatment, 3 months follow up, 6 months follow up.
  Interview administration of the CAPS by independent assessor captures current (past month) and lifetime symptoms and diagnosis of Post-Traumatic Stress Disorder (PTSD).

SECONDARY OUTCOMES:
Change in mental and physical functioning from baseline on the Health Related Quality of Life (SF36) to post-treatment, 3 months, and 6 months later. | Baseline, post-treatment, 3-month follow up, 6-month follow up
  Self-report questionnaire measures 8 life-functioning scales summarized by two content scales--Mental and Physical functioning.
Change in quality of life from baseline on the Quality of Life Inventory (QOLI) to post-treatment, 3 months, and 6 months later. | Baseline, post-treatment, 3-month follow up, 6-month follow up
  QOLI is a self-report questionnaire measuring overall quality of life across 16 domains.
Change in PTSD from baseline to points during treatment with the PTSD Symptom Checklist (PCL). | Baseline, after each treatment block (every 5 weeks), post-treatment
  The PCL is a self-report questionnaire measuring 17 PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Diane T Castillo, Ph.D., Principal Investigator — New Mexico VA Healthcare System
Locations (1):
- New Mexico VA Health Care System, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Foa EB, Rothbaum BO, Riggs DS, Murdock TB. Treatment of posttraumatic stress disorder in rape victims: a comparison between cognitive-behavioral procedures and counseling. J Consult Clin Psychol. 1991 Oct;59(5):715-23. doi: 10.1037//0022-006x.59.5.715. PMID 1955605
- [Background] Schnurr PP, Friedman MJ, Engel CC, Foa EB, Shea MT, Chow BK, Resick PA, Thurston V, Orsillo SM, Haug R, Turner C, Bernardy N. Cognitive behavioral therapy for posttraumatic stress disorder in women: a randomized controlled trial. JAMA. 2007 Feb 28;297(8):820-30. doi: 10.1001/jama.297.8.820. PMID 17327524
- [Background] Keane TM , Fairbank JA , Caddell JM , Zimering RT : Implosive (flooding) therapy reduces symptoms of PTSD in Vietnam combat Veterans . Behav Ther 1989 ; 20: 245 - 60 .
- [Background] Resick PA, Schnicke MK. Cognitive processing therapy for sexual assault victims. J Consult Clin Psychol. 1992 Oct;60(5):748-56. doi: 10.1037//0022-006x.60.5.748. PMID 1401390
- [Background] Cahill SP, Rothbaum BO, Resick P, & Follette VM. Cognitive-behavioral therapy for adults. In E. B. Foa, T. M. Keane, M. J. Friedman, & J. A. Cohen (Eds.), Effective treatments for PTSD: Practice Guidelines from the International Society for Traumatic Stress Studies (pp. 139-222). New York: The Guildford Press, 2009.
- [Background] Garrick J : Efficacy of PTSD treatment in the VA . VHSJ 2000 : 5: 15-21 .
- [Background] Schnurr PP, Friedman MJ, Foy DW, Shea MT, Hsieh FY, Lavori PW, Glynn SM, Wattenberg M, Bernardy NC. Randomized trial of trauma-focused group therapy for posttraumatic stress disorder: results from a department of veterans affairs cooperative study. Arch Gen Psychiatry. 2003 May;60(5):481-9. doi: 10.1001/archpsyc.60.5.481. PMID 12742869
- [Background] Castillo DT : Systematic outpatient treatment of sexual trauma in women: Application of cognitive and behavioral protocols . Cogn Behav Pract 2004 : 11: 352 - 65 .
- [Background] Castillo DT, C' de Baca J, Qualls C, Bornovalova MA. Group exposure therapy treatment for post-traumatic stress disorder in female veterans. Mil Med. 2012 Dec;177(12):1486-91. doi: 10.7205/milmed-d-12-00186. PMID 23397693